CLINICAL TRIAL: NCT06169410
Title: Evaluation of the Efficacy and Safety of Ramucirumab Combined With Nab-paclitaxel, Lobaplatin, and S-1 in Neoadjuvant and Conversion Therapy for Advanced Gastric Cancer (RNPLS-01)
Brief Title: Ramucirumab Combined With Nab-paclitaxel, Lobaplatin, and S-1 in Neoadjuvant Transformation Therapy for Advanced Gastric Cancer
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yang Jianjun, PhD (Other)
Responsible Party: Sponsor-Investigator, Yang Jianjun, PhD, Professor from Xijing Hospital, Xijing Hospital
Organization: Xijing Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RNPLS-01
Record Dates: First submitted 2023-11-19; First posted 2023-12-13 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Advanced Gastric Cancer
Keywords: Ramucirumab; nab-Paclitaxel; lobaplatin; S-1; advanced gastric cancer
MeSH Terms: interventions — 130-nm albumin-bound paclitaxel; lobaplatin; Ramucirumab; S 1 (combination)

STUDY DESIGN:
Masking Description: Although this trial was designed as open label, other independent researchers who conducted the imaging evaluation will be in a blinded state in the imaging evaluation phase for reducing the evaluator bias.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ramucirumab combined with lobaplatin, S-1 and nab-paclitaxel (Experimental): Patients will be given ramucirumab (8mg/kg), lobaplatin (30 mg/m2) and nab-paclitaxel (100mg/m2) by intravenous drip on the first day of each cycle, 3 weeks a cycle, together with oral S-1 (patients with a body surface area less than 1.25 m2, will give 40 mg each time; patients with a body surface area between 1.25 and 1.5 m2; will give 50 mg each time; patients with a body surface area greater than 1.5 m2, will give 60 mg each time), 2 weeks on and 1 week off.
  Interventions: Drug: nab-paclitaxel, lobaplatin, and S-1 combined with ramucirumab; Drug: nab-paclitaxel, lobaplatin, and S-1
- lobaplatin combined with S-1 and nab-paclitaxel (Active Comparator): Patients will be given lobaplatin (30 mg/m2) and nab-paclitaxel (100mg/m2) by intravenous drip on the first day of each cycle, 3 weeks a cycle, together with oral S-1 (patients with a body surface area less than 1.25 m2, will give 40 mg each time; patients with a body surface area between 1.25 and 1.5 m2; will give 50 mg each time; patients with a body surface area greater than 1.5 m2, will give 60 mg each time), 2 weeks on and 1 week off.
  Interventions: Drug: nab-paclitaxel, lobaplatin, and S-1

INTERVENTIONS:
Drug: nab-paclitaxel, lobaplatin, and S-1 combined with ramucirumab — Patients in Experimental group will be given ramucirumab (8mg/kg) by intravenous drip on the first day of each cycle, 3 weeks a cycle.
  Arms: ramucirumab combined with lobaplatin, S-1 and nab-paclitaxel
Drug: nab-paclitaxel, lobaplatin, and S-1 — Patients will be given lobaplatin (30 mg/m2) and nab-paclitaxel (100mg/m2) by intravenous drip on the first day of each cycle, 3 weeks a cycle, together with oral S-1 (patients with a body surface area less than 1.25 m2, will give 40 mg each time. Patients with a body surface area between 1.25 and 1.5 m2; will give 50 mg each time; patients with a body surface area greater than 1.5 m2, will give 60 mg each time), 2 weeks on and 1 week off.

SUMMARY:
Abstract Objective: Ramucirumab is a VEGFR2 antagonist. The aim of this trial is to evaluate the efficacy and safety of ramucirumab combined with nab-paclitaxel, lobaplatin and S-1 in neoadjuvant and conversion therapy for advanced gastric cancer.

Methods and analysis: This study is a prospective single-center, randomized controlled and open label clinical study containing two cohorts with 140 patients of advanced gastric cancer (Cohort A n=70; Cohort B n=70). The main efficacy indicator is pathological complete response (pCR) of the cancer after neoadjuvant or conversion therapy. The secondary efficacy indicators are R0 resection rate after neoadjuvant or conversion therapy, the incidence of adverse events (AE), progression-free survival (PFS), overall survival (OS), objective response rate (ORR), total response rate and total response time, disease control rate (DCR) and duration of overall response (DOR).

Ethics: Ethics approval has been obtained from the Ethics Committee at the First Affiliated Hospital (Xijing Hospital) of Air force Military Medical University (KY20232220-F-1).

ELIGIBILITY:
Inclusion Criteria:

Cohort A: Patients are diagnosed with locally advanced gastric or gastroesophageal junction adenocarcinoma by cytology or histopathology and in need of preoperative neoadjuvant therapy to reduce recurrence and metastasis rates; Cohort B: Patients with advanced gastric cancer who have undergone surgery after neoadjuvant chemotherapy with previously used nab-paclitaxel, lobaplatin and S-1.

Patients are adults aged 18-75 years with an Eastern Cooperative Oncology Group(ECOG) performance status score less than or equals to 1.

Have not received anti-tumor treatment (such as surgery, radiotherapy, chemotherapy, targeted therapy, immunotherapy) .

Functions of the major organs and bone marrow meet the following criteria within 7 days before treatment: hemoglobin ≥ 80g/L, absolute neutrophil count ≥ 1.5 × 109/L, platelet (PLT) ≥ 100× 109/L, without blood transfusion within 14 days, total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal (ULN). Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5x ULN or if complicated with liver metastasis then ALT and AST ≤ 5x ULN, serum creatinine ≤ 1.5x ULN or creatinine clearance ≥ 50mL/min or urinary protein<2+, activated partial thromboplastin time (APTT) and international standardized ratio (INR)≤1.5×ULN.

Expected lifespan ≥ 6 months. The patients are able and willing to provide written informed consent to participate in the study.

Exclusion Criteria:

Patients who have previously suffered from other malignant tumors, except for cured skin basal cell carcinoma and cervical carcinoma in situ.

HER-2 positive patients who are willing to receive Herceptin treatment. Women who are pregnant or lactating or in the reproductive period and have not taken effective contraceptive measures, or those who have fertility requirements during the research period.

Patients with serious and uncontrolled internal diseases and infections or with chronic bowel disease or short bowel syndrome.

Patients with major organ failure, such as compensatory heart, lung, liver, and kidney failure as well as severe metabolic abnormalities in liver and kidney which affects normal drug metabolism.

Patients with a clear tendency for gastrointestinal bleeding and/or abnormal coagulation function (INR>1.5)under researchers evaluation.

hepatitis B virus or hepatitis C virus in active phase Patients with peripheral neuropathy neoadjuvant chemotherapy(NCT)-CTCAE ≥ Level 2.

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-12-30 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
pCR | 48 months
  pathological complete response

SECONDARY OUTCOMES:
R0 resection rate | 48 months
  R0 resection rate after neoadjuvant or conversion therapy
AE | 48 months
  the incidence of adverse events (AE)
PFS | 48 months
  progression-free survival (PFS)
OS | 48 months
  overall survival (OS)
ORR | 48 months
  objective response rate (ORR)
total response rate | 48 months
  total response rate
DCR | 48 months
  disease control rate (DCR)
DOR | 48 months
  duration of overall response (DOR)
total response time | 48 months
  total response time

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of the Air Force Medical University, Xi'an, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wang J, Xu G, Liu S, Ma Y, Wang S, Li M, Zhao Y, Wang H, Wang Y, Peng C, Huo H, Li H, Ji G, Yang J. Evaluation of the efficacy and safety of ramucirumab combined with nab-paclitaxel, lobaplatin, and S-1 in neoadjuvant and conversion therapy for advanced gastric cancer: A study protocol of prospective single-center, randomized controlled and open label clinical trial (RNPLS-01). Heliyon. 2024 Apr 9;10(8):e29485. doi: 10.1016/j.heliyon.2024.e29485. eCollection 2024 Apr 30. PMID 38660276